CLINICAL TRIAL: NCT01211158
Title: A Randomized Double-blind Trial to Evaluate Ketamine-propofol Combination vs. Propofol Alone for Procedural Sedation and Analgesia in the Emergency Department.
Brief Title: Ketofol vs Propofol for Emergency Department Procedural Sedation and Analgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lions Gate Hospital (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Gary Andolfatto, Clinical Assistant Professor, Department of Emergency Medicine, University of British Columbia, Lions Gate Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: gandolfatto
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Emergency Department Procedural Sedation; Fracture Reduction; Abscess Incision and Drainage; Electrical Cardioversion
Keywords: emergency department; procedural sedation; ketofol; ketamine; propofol; conscious sedation
MeSH Terms: conditions — Emergencies | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol alone (Active Comparator): Patients receiving propofol alone.
  Interventions: Drug: Propofol alone
- Ketofol (Active Comparator): 0.375 mg/kg each of ketamine and propofol (mixed in the same syringe) as an initial bolus and 0.188 mg/kg each of ketamine and propofol as necessary until reaching deep sedation (Ramsay score = 5 or greater).
  Interventions: Drug: Ketofol

INTERVENTIONS:
Drug: Ketofol — Syringes containing ketofol (mixed propofol-ketamine) will contain propofol 5mg/ml and ketamine 5 mg/ml. Patients will receive an initial intravenous dose of 0.075 millilitres per kilogram of pre-prepared medication. Patients in the propofol-ketamine group will receive 0.375 mg/kg each of ketamine and propofol as an initial bolus and 0.188 mg/kg each of ketamine and propofol as necessary until reaching deep sedation (Ramsay score = 5 or greater).
  Other Names: single-syringe ketamine-propofol 1:1 combination
  Arms: Ketofol
Drug: Propofol alone — Propofol-only syringes will contain propofol 10 mg/ml. Patients in each group will receive an initial intravenous dose of 0.075 millilitres per kilogram of pre-prepared medication (0.75 mg/kg). One minute after the initial dose of sedative, and every minute thereafter, the attending physician will assess the patient's level of sedation using the Ramsay Sedation Scale (RSS). If the attending physician determines the level of sedation to be inadequate (RSS<5), additional study drug will be administered at a dose of 0.0375 millilitres per kilogram (0.375 mg/kg) every minute until deep sedation is achieved (RSS=5 or greater).
  Other Names: Diprivan
  Arms: Propofol alone

SUMMARY:
When patients come to the Emergency Department with injuries and infections they often need to have painful procedures performed that are essential to allowing them to recover. To accomplish this, doctors often use "procedural sedation". This involves giving medications through an intravenous line in order to relieve the patient's pain and to make them drowsy while the painful procedure is being performed. This allows the medical staff to perform necessary procedures to patients without causing pain and anguish.

There are several types of medications and combinations of medications that are used for procedural sedation. Each medication has its advantages and its disadvantages. Consequently, research is necessary to determine which medication or combination of medications is the most effective and the safest. This study will compare the use of one drug (Propofol) versus the use of a combination of Propofol with another drug (Ketamine). Both of these drugs are already used for procedural sedations in the emergency department but it is not known which of them is the best or the safest.

The investigators believe that the combination of ketamine and propofol together will work as good or better than propofol alone and be a safer option as well. Propofol is a well known sedative that is used in many emergency departments and the clinical experience with it has been very good because it acts quickly and wears off quickly. However, propofol is not a good pain-killer and it can also cause patients to stop breathing. This is why monitoring a patient's breathing and vital signs is essential for any procedural sedation. It is known that ketamine is a good pain-killer and helps patients to maintain their breathing. Doctors sometimes use ketamine alone for procedural sedation but patients take a very long time to wake up when ketamine only is used.

Thus, the investigators think that by combining ketamine with propofol the investigators can perform painful procedures using procedural sedation without causing patients to stop breathing as often as with propofol alone. Also, the ketamine the investigators use will help treat their pain and make them more comfortable.

The investigators plan to enroll 284 patients over the course of about one year. The primary outcome of adverse respiratory events, as well as the secondary outcomes will be assessed during the course of the sedation and recovery period, approximately one hour. Quality of life score and pain will be assessed by telephone interview 3 days after the procedure.

DETAILED DESCRIPTION:
Procedural sedation and analgesia (PSA) for painful procedures is the standard of care in emergency medicine.

The ideal PSA agent should be safe, easy to administer, provide analgesia and amnesia with rapid onset, quick recovery and a minimum of adverse effects. A variety of medications have been studied for procedural sedation but no single medication currently used meets all of these criteria. Two medications that are well known and often used for procedural sedation are propofol and ketamine. Both medications have been shown to be highly effective but each has important limitations in emergency practice. Propofol is known to cause respiratory depression, apnea, and hypotension in a dose-dependent fashion. Ketamine displays a longer recovery time than propofol and patients receiving ketamine sedation are prone to vomiting and unpleasant emergence reactions. The use of ketamine and propofol in combination is theoretically compelling as the sedative effects of propofol should logically balance the nauseant and psychomimetic effects of ketamine while the ability to achieve deep sedation with lower doses of ketamine should logically permit for a shorter physiologic recovery time compared ketamine alone. As well, ketamine provides an analgesic effect that is absent with propofol and has been shown to be safer than using opioid analgesia such as fentanyl when considering airway events. This study seeks to evaluate a ketamine-propofol combination that potentially provides effective procedural sedation and analgesia while exposing patients to less risks associated with respiratory depression as the differential effects of ketamine and propofol may lead to fewer adverse events than either medication used alone.

Propofol is a nonopioid, nonbarbiturate, sedative-hypnotic agent whose desirable properties include its rapid onset, short duration of action, and reliability in producing sedation. It also acts an anti-emetic but has no analgesic properties. Adverse effects include dose-related cardiovascular and respiratory depression and bradycardia. This dose-dependent respiratory depression, apnea and hypotension may present barriers to the widespread clinical utility of propofol. In addition, the lack of an analgesic effect may necessitate the use of other agents to provide pain relief during procedural sedation. The use of opioid analgesia in conjunction with propofol sedation is well known to increase the risk of adverse airway events.

Ketamine is an agent classified as a dissociative sedative and is known to provide efficacious and safe procedural sedation with the preservation of airway reflexes and respiratory drive. The use of ketamine for severe acute pain in the emergency department has been shown to decrease opioid requirements in trauma patients as well as reduce the pain of propofol injection. During deep sedation with propofol, the use of sub-dissociative ketamine for analgesia during emergency department procedural sedation results in fewer adverse airway events than does fentanyl. The main limitations of the use of ketamine alone for procedural sedation is its longer recovery time and the incidence of dysphoric emergence reactions, especially in adults.

Ketamine-propofol combination has been used successfully and safely for a variety of purposes, including gynecological and ophthalmological procedures, sedation for spinal anesthesia, and cardiovascular procedures in both adults and children. Ketamine and propofol mixed in the same syringe has been shown to be safe and effective in both the operating room and in the office setting. Combining ketamine with propofol appears to provide anesthetic synergy with a widened therapeutic index, permitting the induction of anesthesia and sedation at doses less likely to lead to respiratory depression. Thus, the combination of ketamine and propofol has received interest as an emergency department procedural sedation regimen that allows the provision of PSA using drug doses lower than typically required for each agent alone potentially resulting in fewer adverse effects and shorter recovery times. Propofol is a potent sedative and with anti-nauseant properties and is thought to likely mitigate the problematic adverse psychomimetic and nauseant effects of ketamine. Ketamine and propofol are known to be physically and chemically stable when mixed in polypropylene syringes and the mixture displays stable respiratory and hemodynamic parameters in healthy patients during general anesthesia. The use of ketamine and propofol in combination in the ED is limited. A pilot study of 20 children showed that ketamine and propofol administered from separate syringes to ED patients resulted in reliable deep sedation with few adverse effects. Prospective ED case series in children and in adults have shown that ketamine and propofol mixed in a single syringe in a 1:1 ratio (so called "ketofol") appears to be an effective ED PSA agent that is well tolerated and appears safe. To date, there has not been any randomized trial comparing single-syringe ketofol with other known ED PSA agents, thus the theoretical advantages of ketamine-propofol combination (ketofol) are not yet definitively known.

Methodology Experimental Design: This study will be a prospective, double-blind, randomized clinical trial. A systematic review of the literature on propofol use in emergency department procedural sedation using explicit criteria was carried out. Trials were selected based on the following criteria: 1) propofol alone was the sedation agent used, 2) At least a 30 minute "washout" period between pre-procedural analgesic use before the commencement of procedural sedation, 3) Propofol used in an intermittent bolus technique, 4) Patients greater than 14 years of age, 5) Study published less than 10 years previously, 6) Study performed in the emergency department.

Nine studies were identified totaling 1679 patients. These were reviewed with respect to reported airway events based on the Quebec Criteria definitions for airway events. The composite adverse airway event from these studies was 21% (95% CI 19.05% to 22.95%).

The composite Quebec Criteria adverse event rate for studies of ketamine-propofol sedation was then determined from the available literature. Three studies were identified with a total enrollment of 166 patients. Airway event data from a prospective case series (n=328) performed at LGH was also included. The pooled results yielded a composite adverse airway event rate of 8% (95% CI 5.87% to 10.73%).

Based on these data (21% event rate in the propofol arm, 8% anticipated event rate in the ketamine-propofol arm), 129 subjects would be needed in each group (total 258 subjects) to have 80% power to detect a difference of this magnitude or greater (alpha 0.05, two-sided calculation). An additional 10% enrollment will be added to the total enrollment to offset potential drop-outs, resulting in a total sample size of 284 subjects (142 in each arm). Written, informed consent will be obtained from all patients or from a parent/guardian in those under the age of 18 years.

Enrollment Projection: The emergency department at Lions Gate Hospital presently performs an average of 55 procedural sedations per month. Assuming a 50% enrollment rate (based on local enrollment experience in other ED randomized trials), it would be expected that full study enrollment would occur within 12 months.

All patients will receive pre-procedural analgesia at the discretion of the treating physician. For entry into the study there will be a minimum 30-minute "washout" period between analgesic use and the commencement of the procedural sedation. Sealed envelopes containing a randomized assignment to either propofol-alone or ketamine-propofol will be prepared using a web-based random number generator. Block randomization will be done (random block sizes) to ensure an approximate of allocations between the two arms of he study throughout enrollment, thus maximizing statistical power if any unanticipated events lead to trial termination prior to complete enrollment. Data, including crossovers or contamination (both of which are exceedingly unlikely) will be analysed on an Intent to Treat principle.

Identical pre-prepared syringes will contain either propofol-alone or ketamine-propofol mixture, prepared by trained and in-serviced registered nurses. Medications will be overseen by the emergency department clinical pharmacist. To assist in blinding, patients will wear reflective sunglasses in order to obscure eye movements (nystagmus - a known effect of ketamine) from the study investigators.

All sedations will be performed under continuous cardiorespiratory monitoring as directed under the Vancouver Coastal Health Authority Guidelines for Emergency Department Procedural Sedation and Analgesia. All procedural sedation events will require the attendance of a certified emergency physician, registered nurse, and respiratory therapist. Vital signs including heart rate, respiratory rate, oxygen saturation, and end-tidal carbon dioxide will be monitored continuously and recorded every 2 minutes. Blood pressure will be recorded every 4 minutes.

A separate, standardized data sheet will be used to collect the time of study drug administration, time of procedure start, time of procedure completion, and time of physiologic recovery. Recovery will be assessed after completion of the procedure by the use of a modified Aldrete Scale every 2 minutes until full recovery, defined as a minimum cumulative score of 8. The attending physician will be asked to document any complications that occurred during the procedure and if any interventions were necessary. The nurse caring for the patient will also be asked to record any adverse events occurring during the recovery phase. To evaluate the success of study blinding, at the conclusion of each sedation the attending physician and nurse will be asked to independently guess whether the patient in question received propofol-only or ketamine-propofol. Primary and secondary outcomes will be assessed during the course of the sedation procedure and recovery, less than one hour in the vast majority of cases. Quality of Life and pain scores will be assessed by telephone interview 72 hours after the sedation procedure.

Analysis: Statistical consultation prior to the study launch was obtained through the VCHRI Centre for Clinical Epidemiology and Evaluation (C2E2).

Analysis of primary outcome:

The number proportion of patients suffering a respiratory AE will be reported by treatment group. A 95% CI for the difference between treatment groups will be determined. The equality of the two proportions will be tested using Fisher's exact test.

Analysis of secondary outcomes:

Quality of sedation. The number and proportion of patients with a RSS < 5 during the procedure, or requiring further sedation at any time during the procedure will be reported for each treatment group. The equality of the two proportions will be tested using Fisher's exact test. For all other secondary outcomes only descriptive analyses are planned.

Analysis of safety outcomes:

Frequencies and percentages of complications and adverse events (excluding respiratory) by treatment group will be reported with 95% CI's.

Interim Analyses:

There are no planned interim analyses for either efficacy or safety.

The Mann-Whitney test will be used to compare differences in satisfaction levels (measured on an ordinal scale) between groups.

A p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age 14 years or greater
* deemed to require emergency department procedural sedation by the attending physician

Exclusion Criteria:

* unable to give informed consent
* hemodynamic instability
* pregnancy
* known allergy to either study medication

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number and proportion of patients experiencing a respiratory adverse event as described by the Quebec Criteria | 1 hour
  Oxygen desaturation, central apnea, partial upper airway obstruction, complete upper airway obstruction, laryngospasm, clinically apparent pulmonary aspiration.

SECONDARY OUTCOMES:
Quality of sedation | During procedure - average time 5 - 10 minutes
  Number of patients maintaing Ramsay Sedation Score (RSS) of 5 or greater throughout the procedure; Number of patients requiring repeat dosing of medication to maintain RSS 5 or greater.
Sedation complications | During procedure and recovery period and before discharge - average time 1-2 hours
  unplanned reversal agent use, unexpected hospital admission due to sedation
Post-procedural patient comfort | 72 hours post sedation
  SF-8 Quality of Life Survey (QualityMetric Inc., Lincoln, RI) and pain-score assessment (10-point Likert scale).
Hypotension | During sedation and recovery - average time 30-45 minutes
  Number of patients experiencing drop in systolic blood pressure below 90 mmHg and requiring intervention such as intravenous fluid bolus or vasopressors.
Recovery agitation requiring treatment | During recovery period - average time 30 - 45 minutes
  Number of patients requiring intervention (medication or restraint) for recovery agitation
Bradycardia | During procedure and recovery period - average time 30-45 minutes
  Number of patients with heart rate less than 60 beats per minute requiring intervention.
Muscular rigidity | during procedure - average time 5 - 10 minutes
  Number of patient experiencing muscular rigidity interfering with the procedure.
Vomiting | 1 hour
  vomiting or retching during procedure and recovery period
Recovery agitation not requiring treatment | 1 hour
  Patients with apparent recovery agitation but not requiring administration of medication
Induction time | 1 - 15 min
  Time and number of medication doses required to achieve RSS 5 or greater.
Procedural agitation | 1 - 20 min
  as judged by the treating physician - patient combativeness, paradoxical response to medication, reactivity to painful manipulation - interfering with procedure
Sedation Efficacy | 1 hour
  1) Patient does not have unpleasant recall of the procedure; 2) Patient did not experience an adverse event resulting in abandonment of the procedure, a permanent complication, prolonged ED observation, or unplanned admission to hospital; 3) Patient did not actively resist or require physical restraint for completion of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Andolfatto, MD, Principal Investigator — Lions Gate Hospital, University of British Columbia Department of Emergency Medicine
Locations (1):
- Lions Gate Hospital, North Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bhatt M, Kennedy RM, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM, Roback MG; Consensus Panel on Sedation Research of Pediatric Emergency Research Canada (PERC) and the Pediatric Emergency Care Applied Research Network (PECARN). Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009 Apr;53(4):426-435.e4. doi: 10.1016/j.annemergmed.2008.09.030. Epub 2008 Nov 20. PMID 19026467
- [Background] Messenger DW, Murray HE, Dungey PE, van Vlymen J, Sivilotti ML. Subdissociative-dose ketamine versus fentanyl for analgesia during propofol procedural sedation: a randomized clinical trial. Acad Emerg Med. 2008 Oct;15(10):877-86. doi: 10.1111/j.1553-2712.2008.00219.x. Epub 2008 Aug 27. PMID 18754820
- [Background] Miner JR, Gray RO, Stephens D, Biros MH. Randomized clinical trial of propofol with and without alfentanil for deep procedural sedation in the emergency department. Acad Emerg Med. 2009 Sep;16(9):825-34. doi: 10.1111/j.1553-2712.2009.00487.x. PMID 19845550
- [Background] Miner JR. The surgical stress response, preemptive analgesia, and procedural sedation in the emergency department. Acad Emerg Med. 2008 Oct;15(10):955-8. doi: 10.1111/j.1553-2712.2008.00249.x. No abstract available. PMID 18851717
- [Background] Arora S. Combining ketamine and propofol ("ketofol") for emergency department procedural sedation and analgesia: a review. West J Emerg Med. 2008 Jan;9(1):20-3. No abstract available. PMID 19561698
- [Background] Sharieff GQ, Trocinski DR, Kanegaye JT, Fisher B, Harley JR. Ketamine-propofol combination sedation for fracture reduction in the pediatric emergency department. Pediatr Emerg Care. 2007 Dec;23(12):881-4. doi: 10.1097/pec.0b013e31815c9df6. PMID 18091596
- [Result] Andolfatto G, Willman E. A prospective case series of pediatric procedural sedation and analgesia in the emergency department using single-syringe ketamine-propofol combination (ketofol). Acad Emerg Med. 2010 Feb;17(2):194-201. doi: 10.1111/j.1553-2712.2009.00646.x. PMID 20370749
- [Result] Willman EV, Andolfatto G. A prospective evaluation of "ketofol" (ketamine/propofol combination) for procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2007 Jan;49(1):23-30. doi: 10.1016/j.annemergmed.2006.08.002. Epub 2006 Oct 23. PMID 17059854